CLINICAL TRIAL: NCT03359616
Title: Transanal Versus Laparoscopic Total Mesorectal Excision for Mid And Low Rectal Cancer in China (TLTME): a Single-center Randomized Clinical Trial
Brief Title: Transanal Versus Laparoscopic Total Mesorectal Excision For Rectal Cancer
Acronym: TLTME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MISC-TaTME
Record Dates: First submitted 2017-11-26; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Rectal Cancer; Surgery
Keywords: rectal cancer; laparoscopic surgery; total mesorectal excision; transanal surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transanal total mesorectal excision (Experimental): Transanally, the rectum is mobilized through the mesorectal plane according to the TME principles, assisted by the transanal surgical platform (Transanally curable surgical resection).
  Interventions: Procedure: Transanally curable surgical resection
- laparoscopic total mesorectal excision (Active Comparator): By standard laparoscopic techniques, the rectal cancer will be resected by the conventional laparoscopic TME (LaTME).
  Interventions: Procedure: Laparoscopic total mesorectal excision

INTERVENTIONS:
Procedure: Transanally curable surgical resection — Transanally, the rectal cancer will be mobilized with oncological principle of total mesorectal excision
  Arms: transanal total mesorectal excision
Procedure: Laparoscopic total mesorectal excision — Conventionally by laparoscopic surgery, the rectal cancer will be mobilized with oncological principle of total mesorectal excision
  Arms: laparoscopic total mesorectal excision

SUMMARY:
Total mesorectal excision (TME) has been prevailingly accepted as a crucial surgical intervention within the latest oncological therapeutic regime for mid-low rectal cancer. However, surgical dissection under the restricted pelvic anatomical structure, added by obesity and many other general factors, remains challenging for classical open and laparoscopic patterns, particularly in male cases. The introduction of transanal total mesorectal excision (TaTME) offers an optimal pattern for the surgical resection of mid-low rectal cancer, circumventing the conventional anatomical limits while bringing forward considerable advantages by direct dissection. Noteworthy, the surgical techniques of TaTME is initially established, with the mortality/morbidity and the oncological safety unverified. The studies that focus on the comparison between TaTME and laparoscopic TME (LaTME) remain sparse. Therefore, the features of TaTME, both in short and long terms, await further consolidation by clinical trials. Herein, this single centered, interventional study protocol is established to collect initial clinical data on both the safety and efficacy of the TaTME in comparison with LaTME in East Chinese patients with mid-low rectal cancer.

DETAILED DESCRIPTION:
Background: Transanal total mesorectal excision (TaTME) is increasingly accepted as one of the alternative patterns for the resectable rectal cancer worldwide since its first appearance. For mid-low rectal cancer, TaTME features superior viewpoints and direct access to mobilize the primary lesion without the pelvic anatomic limits. Therefore, the matured TaTME technique could deliver satisfactory clinic outcomes in both surgical and oncological senses. However, the studies that designed to compare the feasibility and repeatability of TaTME with conventional laparoscopic total mesorectal excision (LaTME) remain sparse and limited.

Study Objective: Evaluation of short-term mortality and morbidity, long term overall survival and disease-free survival as well as quality of life in rectal cancer patients in East China.

Study Design: This study is a prospective, single-center, randomized clinical trial with a central monitored electronic data processing system. Corresponding randomization, data collection and comparative analysis will be conducted based on the research group discussion. According to the non-inferiority principle, the power is 80% and the α is 0.05 with 10% margin delta (δ). Total patients will be 258, with 129 in each group given 10% lost in follow-up.

Study Endpoints: The primary outcomes measures will be the Disease-free survival (3-years). The secondary outcomes measures will be overall survival (3-years), mesorectal completeness (the quality of the TME specimen, complete, near complete, incomplete), positive circumferential resection margin (CRM), number of retrieved lymph nodes, morbidity rate, mortality rate.

ELIGIBILITY:
Inclusion Criteria:

1. Rectal adenocarcinoma validated by pathologists, pathological estimated stage II-III;
2. Mid and low rectal tumor sites, parameter less than 5cm, below the level of peritoneal reflection and verified by MRI, distance to anus less than 7 cm;
3. Curative rectal cancer surgery;
4. No evidence of distance metastasis lesions;
5. T1-3, N0-2, with or without neoadjuvant therapeutic history;
6. Applied to laparoscopic surgery;
7. Absent of previous malignancy-treated history
8. No gender restriction, age between 18 and 75, Body Mass Index less than 32;
9. Approved by multiple disciplinary teamwork therapeutic group
10. Consent by the patient and the family.

Exclusion Criteria:

1. Mile's surgery is additionally required;
2. Tumor invasion is validated on adjacent organs, such as prostate;
3. Recurrent rectal cancer, require secondary surgical interventions;
4. Previous history of malignant diseases or inflammatory bowel diseases within recent five years;
5. Emergent surgery accompanied by bowel obstruction or intestinal perforation;
6. Previous history of colorectal surgery, unnatural anatomical structure;
7. Contraindication to general anesthesia (class IV or V in American Society of Anesthesiologists (ASA), or Eastern Cooperative Oncology Group (ECOG) score >=2)
8. Pregnant or breast-feeding patients;
9. Mental disorder validated by psychiatrists.
10. Uncontrolled infectious diseases;
11. Participants within other related clinical trials that may influence the conclusion of this trial;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3-years
  3-year DFS

SECONDARY OUTCOMES:
Overall survival (OS) | 3-years
  3-years OS
mesorectal completeness | 3-years
  (the quality of the TME specimen, complete, near complete, incomplete)
positive circumferential resection margin | 3-years
  the rate of positive circumferential resection margin (CRM)
number of retrieved lymph nodes | 3-years
  retrieved lymph nodes
morbidity rate | 3-years
  morbidity rate(number of intr-and post-operative encountered cases)
mortality rate | 3-years
  (number of intr-and post-operative encountered complications)

CONTACTS AND LOCATIONS:
Overall Officials: Minhua Zheng, M.D., PhD., Study Director — MISC, Ruijin Hospital, School of Medicine, Shanghai Jiao Tong University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Motson RW, Whiteford MH, Hompes R, Albert M, Miles WF; Expert Group. Current status of trans-anal total mesorectal excision (TaTME) following the Second International Consensus Conference. Colorectal Dis. 2016 Jan;18(1):13-8. doi: 10.1111/codi.13131. PMID 26400670
- [Background] Bulut O, Levic K, Hesselfeldt P, Bulow S. The outcome of rectal cancer after early salvage TME following TEM compared with primary TME: a case-matched study. Tech Coloproctol. 2014 Jan;18(1):83-4. doi: 10.1007/s10151-013-1083-y. Epub 2013 Nov 6. No abstract available. PMID 24197900
- [Background] Martin-Perez B, Andrade-Ribeiro GD, Hunter L, Atallah S. A systematic review of transanal minimally invasive surgery (TAMIS) from 2010 to 2013. Tech Coloproctol. 2014 Sep;18(9):775-88. doi: 10.1007/s10151-014-1148-6. Epub 2014 May 7. PMID 24848524
- [Result] Fernandez-Hevia M, Delgado S, Castells A, Tasende M, Momblan D, Diaz del Gobbo G, DeLacy B, Balust J, Lacy AM. Transanal total mesorectal excision in rectal cancer: short-term outcomes in comparison with laparoscopic surgery. Ann Surg. 2015 Feb;261(2):221-7. doi: 10.1097/SLA.0000000000000865. PMID 25185463